CLINICAL TRIAL: NCT03448146
Title: A Phase III Single Arm Trial of PTS (Para Toluenesulfonamide Injection) Via Bronchoscopy Intervention Intratumoral Injection in Patients With Central Air Way NSCLC Tumor Severe Obstruction
Brief Title: A Trial of PTS Via Intratumoral Injection in Patients With Central Air Way NSCLC Severe Obstruction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PTS International Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTS302
Record Dates: First submitted 2018-02-11; First posted 2018-02-27 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Nsclc
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 4-toluenesulfonamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Para-Toluenesulfonamide (Experimental): 1. .The dose of PTS injected into multiple points in a single tumor was about 0.1-1.0 mL, and the appropriate specific doses were kept within the tumor without leakage. An appropriate low dose could be given firstly, and the following doses could be adjusted based on the response of patient and the tumor.
  2. . In general, the daily dose of PTS injected into a single tumor was no more than 5mL, and the daily dose of PTS was no more than 10mL for each patient.
  The injection was provided 2-3 times a week, with 2 weeks as a cycle of treatment. No less than 4 times of PTS treatment were recomended for the first cycle of treatment, and for other cycles of treatment, the number of PTS injections could be adjusted appropriately based on the condition of the patient.
  Interventions: Drug: Para-Toluenesulfonamide

INTERVENTIONS:
Drug: Para-Toluenesulfonamide
  Other Names: PTS

SUMMARY:
This trial was to evaluate the efficacy of intratumoral PTS injection in alleviating airway obstruction and dyspnea by improving the percentage of lumen patency of patients with central air way NSCLC tumor severe obstruction.

DETAILED DESCRIPTION:
1. Local intratumoral injection of para toluenesulfonamide (PTS) via bronchoscopy could alleviate airway obstruction for patients with central air way NSCLC tumor severe obstruction, which contributed to the shrinkage of target tumor lesions in a short period, with an objective response rate of 66% and an improvement rate of luminal tumor obstruction of 70% in the end-of-treatment period.
2. Patient's pulmonary function, atelectasis and quality of life were improved significantly after treatment, indicating that PTS treatment cuold relieve the symptoms of air way obstruction and provide clinical benefits to the patients.
3. Adverse events were mainly blood streaked sputum, injection site haemorrhage, cough, pyrexia and oropharyngeal pain, without reporting of potential risks. Common study drug related adverse events included injection site haemorrhage, cough, and blood streaked sputum and oropharyngeal pain. The multi-center clinical study conducted strictly in accordance with Standard Operation Procedures for the Use of a Standard Bronchoscope in Local Intratumoral PTS Injection showed that PTS had good safety and tolerability and that the procedural risks of intratumoral PTS injection via bronchoscopy could be controlled.
4. The advantages of PTS for treatment of airway lung cancer obstruction included significant efficacy, good safety, large applicable population; relatively simple equipment conditions and operation, thus it could be spread easily. PTS is also expected to be used in the treatment of central lung cancer with acute airway obstruction in combination with other treatments (such as stent implantation), which provides a new drug treatment to patients with airway lung cancer obstruction. PTS can complement with other treatments, which is expected to improve the treatment efficacy significantly.

ELIGIBILITY:
Inclusion Criteria:

* Male or female inpatients, aged 18 to 83 years old.
* Patients with central air way non-small cell lung cancer (NSCLC) severe obstruction; definition of severe airway obstruction: ≥1/2 trachea is obstructed by tumor; and/or block ≥2/3 of primary bronchi, right and middle bronchi. And the longest diameter of the lesion > 0.5 cm.
* Pathologically confirmed lung cancer.
* Patients with tracheal tumor lesions suitable for local intratumoral injection via fibro-bronchoscopy.
* At least one measurable lesion that could be evaluated by imaging examination (bronchoscopy, CT, MRI or X-ray etc.) according to the Response Evaluation Criteria in Solid Tumors.
* Blood platelet count ≥ 100,000/mm3.
* Subjects who were able to understand and comply with the trial protocol and give written consent.

Exclusion Criteria:

* Brain metastases.
* History of cardiovascular diseases, including congestive heart failure > New York Heart Association (NYHA) Grade II. Patients with unstable angina pectoris (angina pectoris symptoms at rest), recent angina pectoris (occurred in the recent 3 months) or with myocardial infarction in recent 6 months must be excluded.
* Severe infections or dysbolism.
* Poor hepatic functional reserve or severe hepatocirrhosis, with abnormal blood coagulation indicators.
* Poor general conditions or cachexia.
* The target lesion had been treated with radiotherapy within 6 months.
* Pregnant or breast-feeding woman.
* Known hypersensitivity to PTS or related compounds.
* Lung cancer lesions not suitable for local treatment.
* Any other reason deemed reasonable by the investigator.

Ages: 18 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 30 days after the last treatment
  The objective response rate of target lesions in patients with central air way NSCLC tumor severe obstruction after PTS treatment were evaluated based on measurement results of CT and bronchoscopy.
Improvement rate of luminal obstructions | 30 days after the last treatment
  The improvement rate of luminal obstructions in patients with central air way NSCLC tumor severe obstruction after PTS treatment were evaluated based on measurement results of CT and bronchoscopy.

SECONDARY OUTCOMES:
Change in FVC | 30 days after the last treatment
  Changes in Forced Vital Capacity (FVC)
Change in FEV1/FVC | 30 days after the last treatment
  Changes in Forced Expiratory Volume in One Second (FEV1)/Forced Vital Capacity (FVC)
Change in BDI score | 30 days after the last treatment
  Changes in Baseline Dyspnea Index (BDI) score. The BDI provides a multidimensional measurement of dyspnea based on 3 domains: functional impairment, magnitude of task and magnitude of effort that evoke dyspnea in activities of daily living, in symptomatic individuals. Rated in five grades from 0 to 4 for each domain. Ranging from 0 to 12. The lower the score, the worse the severity of dyspnea.
Change in pleural effusion | 30 days after the last treatment
  Changes in pleural effusion
Change in ECOG performance status | 30 days after the last treatment
  Changes in Eastern Cooperative Oncology Group (ECOG) performance status
Change in QOL score | 30 days after the last treatment
  Changes in Quality of Life (QOL) score. Quality of life (QOL) was evaluated based on the subject's answers in Functional Assessment of Cancer Therapy-Lung Cancer Subscale (FACT-LCS) questionnaire, version 4. Symptoms of lung cancer were evaluated according to the completed Lung Cancer Subscale (LCS). The FACT-LCS, version 4 is a patient completed questionnaire consisting 36 items that assesses health related quality of life (HRQL) in lung cancer patients. The FACT-LCS, version 4 consists of the 27-item FACT-G assessing generic HRQL concerns and 9-item Lung Cancer Subscale assessing disease-specific issues. Instrument scoring yields a range from 0 to 144 with higher scores representing better patient status.
Duration of response (DOR) of target lesion | 30 days after the last treatment
  Duration of response (DOR) of target lesion

CONTACTS AND LOCATIONS:
Overall Officials: Nan Shan Zhong, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, China

REFERENCES:
- [Result] Li SY, Li Q, Guan WJ, Huang J, Yang HP, Wu GM, Jin FG, Hu CP, Chen LA, Xu GL, Liu SZ, Wu CG, Han BH, Xiang Y, Zhao JP, Wang J, Zhou X, Li HP, Zhong NS. Effects of para-toluenesulfonamide intratumoral injection on non-small cell lung carcinoma with severe central airway obstruction: A multi-center, non-randomized, single-arm, open-label trial. Lung Cancer. 2016 Aug;98:43-50. doi: 10.1016/j.lungcan.2016.05.012. Epub 2016 May 17. PMID 27393505